CLINICAL TRIAL: NCT06850532
Title: Metabolic Health, IGF-1, and Cardiovascular Fitness Responses to High-intensity Interval Training and Moderate-intensity Continuous Training in Combination with Superimposed Neuromuscular Electrical Stimulation
Brief Title: NMES Effects on Substrate Metabolism and IGF-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Nasuh Evrim Acar, ASSISTANT PROFESSOR, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MEUFACULTYOFSPORTSCIENCES_2025; BAP20172TP32576 (Other Grant/Funding Number: Mersin University Scientific Research Projects Commission)
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: The Effects of Neuromuscular Electrical Stimulation on Exercise Performance
MeSH Terms: interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Assessment of baseline anthropometric, demographic and physiological components (Experimental)
  Interventions: Other: IGF-1
- Completion of MICT, MICT+NMES, HIIT, and HIIT+NMES protocols (Experimental)
  Interventions: Other: IGF-1
- Assessment of post-test anthropometric, demographic and physiological components (Experimental)
  Interventions: Other: IGF-1

INTERVENTIONS:
Other: IGF-1 — The effects of NMES coupled with HIIT and MICT on IGF-1 and substrate metabolism has not been studied earlier.

SUMMARY:
The aim of this study is to investigate whether neuromuscular electrostimulation (NMES) training coupled with high-intensity interval training (HIIT) and moderate intensity continuous aerobic training has an effect on the metabolic, cardiovascular and hormonal components compared to respective training protocols without concurrent NMES as a exercise performance enhancement strategy.

ELIGIBILITY:
Inclusion Criteria:

- All participants were healthy with no musculoskeletal injuries and had not participated in lower-body resistance training for six months prior to the study.

Exclusion Criteria:

* Individuals with musculoskeletal injuries and had participated in lower-body resistance training for six months prior to the study has been excluded from the enrollement for the current study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Body composition via Bioelectrical Impedance Analysis (Tanita 418-MA, Japan) | From enrollment to the end of treatment at 8 weeks
  Weight (kg) Total body fat (kg) Total muscle mass (kg) The anthropometric parameters were assessed using Bioelectrical impedance analysis (Tanita 418- MA Japan) before all testing sessions.
Height (cm) via a stadiometer (Holtain Ltd., UK). | From enrollment to the end of treatment at 8 weeks
  Height was measured through a stadiometer in the standing position (Holtain Ltd., Crymych, UK).
Heart rate (bpm) via 12-lead ECG | From enrollment to the end of treatment at 8 weeks
  Heart rate was monitored and recorded throughout baseline and follow-up screenings and all training sessions using 12-lead ECG.
Blood Lactate Concentration (mmol/L) via Lactate Pro 2 analyzer | From enrollment to the end of treatment at 8 weeks
  In each GXT testing session (pre-post), blood samples were collected from the earlobe using a Lactate Pro 2 handheld analyzer (LT-1730, Arkray Inc, Kyoto, Japan) to determine blood lactate concentrations testing session (baseline) and at the end of every two minutes interval.
SERUM INSULIN-LIKE GROWTH FACTOR-1 (IGF-1 ng/mL) | From enrollment to the end of treatment at 8 weeks
  A 5 mL fasting blood sample was drawn from the brachial vein 30 minutes before baseline and follow-up IVO2max tests to measure serum IGF-1 concentrations. Participants rested for 15 minutes before sample collection. Samples were stored at -80 °C and analyzed post-study. Serum IGF-1 levels were measured using Elabscience ELISA kits (detection range: 1.56-100 ng/mL; sensitivity: 0.94 ng/mL) per the manufacturer's instructions.
VO2 - Volume of oxygen (ml/kg/min) VCO2 - Volume of carbon dioxide (ml/kg/min) | From enrollment to the end of treatment at 8 weeks
  During all sessions, VO2 and VCO2 were measured using indirect calorimetry (CareFusion MasterScreen CPX) on an Ergoline Ergoselect 100/200 cycle ergometer. Data was averaged over 15-second intervals during all baseline and follow-up screenings and all training sessions. VO2 and VCO2 were also used to calculate respiratory exchange ratio (RER) during all sessions dividing the VCO2 by VO2.
Energy expenditure (L/min) via indirect calorimetry (CareFusion MasterScreen CPX). | From enrollment to the end of treatment at 8 weeks
  During all sessions, energy expenditure was measured using indirect calorimetry (CareFusion MasterScreen CPX). Data was averaged over 15-second intervals, and substrate utilization was calculated using standard formulas.
  * (GOR)- Oxidation rate of sugar (g/min): 4.585 × VCO2 (L/min) -3.2256 × VO2 (L/min)
    * (GO)- Oxidation amount of sugar (g): Oxidation rate of sugar × Time (min)
      * (FOR)- Fat oxidation rate (g/min): 1.695 × VO2 (L/min) -1.701 × VCO2 (L/min) ④ (FO)- Oxidation amount of fat (g): Oxidation rate of fat × Time (min)
        * (EER)- Energy consumption rate (kcal/min): 3.716 × VO2 (L/min) +1.332 × VCO2 (L/min) ⑥ (EE)- Energy expenditure (kcal): [3.716 × VO2 (L/min) +1.332 × VCO2 (L/min)] × Time (min)
Neuromuscular Electrical Stimulation (NMES) Protocol | From enrollment to the end of treatment at 8 weeks
  The NMES protocol was administered via a four-channel COMPEX SP4.0 (Medicompex SA, Ecublens, Switzerland) electric muscle stimulator using biphasic symmetric rectangular pulsed currents set at 300 μs. COMPEX self-adhesive electrodes were used during muscle stimulation with the COMPEX device. Positive snap electrodes (5×5 cm) with a membrane depolarization that stimulate a 25 cm2 area of the muscle surface were placed on the proximal insertion of vastus medialis and vastus lateralis. The other negative electrode (10×5 cm), measuring 50 cm2 was placed over the femoral triangle, 1-3 cm below the inguinal ligament.
Low-frequency Neuromuscular Electrical Stimulation (NMES) | From enrollment to the end of treatment at 8 weeks
  The low-frequency NMES protocol was administered via a four-channel COMPEX SP4.0 (Medicompex SA, Ecublens, Switzerland) electric muscle stimulator using biphasic symmetric rectangular pulsed currents set at 200 μs. Low-frequency NMES protocol was performed with a duty cycle of 20 seconds on (stimulating) and 20 seconds off (no stimulation) and the pulse width was set at 300 μs (warm-up frequency: 3 Hz, training frequency: 20 Hz, wave: square waveform) to the quadriceps muscle throughout 24 sessions. The duration of training was 30 minutes for sessions 1-6, 36 minutes for sessions 7-12, 42 minutes for sessions 13-18, and 48 minutes for sessions 19-24.
High-frequency Neuromuscular Electrical Stimulation (NMES) | From enrollment to the end of treatment at 8 weeks
  High-frequency NMES protocol was administered via a four-channel COMPEX SP4.0 (Medicompex SA, Ecublens, Switzerland) electric muscle stimulator using biphasic symmetric rectangular pulsed currents set at 300 μs. High-freqeuncy NMES protocol consisted of a 5-minute warm-up (65% VO2max) followed by a 1-minute exercise at 120% VO2max and then a 1-minute "loadless" cycling. This interval was repeated 8 times in sessions 1-6 and progressed to 14 repeated intervals by the 24th session. Participants also received an additional NMES treatment with a duty cycle of 12 seconds on (stimulating) and 8 seconds off (no stimulation) and a pulse width of 300 μs (training frequency: 45-60 Hz, wave: square waveform) to the quadriceps muscle throughout 24 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nevzat Demirci, PhD, Study Director — Mersin University
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF